CLINICAL TRIAL: NCT00742105
Title: A Phase I Study of BGT226, Administered Orally in Adult Patients With Advanced Solid Tumor in Japan
Brief Title: Phase I Study to Determine the Maximum Tolerate Dose (MTD) of BGT226 in Advanced Solid Tumors in Japan
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGT226A1101
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Cancer; Solid Tumor; Advanced Solid Tumor
Keywords: PI3K; mTOR; Advanced solid tumor; Adult
MeSH Terms: conditions — Neoplasms | interventions — 8-(6-methoxypyridin-3-yl)-3-methyl-1-(4-piperazin-1-yl-3-trifluoromethylphenyl)-1,3-dihydroimidazo(4,5-c)quinolin-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BGT226 (Experimental)
  Interventions: Drug: BGT226

INTERVENTIONS:
Drug: BGT226

SUMMARY:
This study will confirm safety and tolerability and determine the MTD of BGT226 in Japanese patients with advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) Performance Status of ≤ 2
* Histologically-confirmed, advanced solid tumors
* Progressive, recurrent unresectable disease
* Age ≥ 20

Exclusion Criteria:

* Hematopoietic:
* No diabetes mellitus or history of gestational diabetes mellitus
* No acute or chronic renal disease
* No acute or chronic liver disease
* No acute or chronic pancreatitis
* No impaired cardiac function or clinically significant cardiac diseases such as ventricular arrhythmia, congestive heart failure, uncontrolled hypertension
* No acute myocardial infarction or unstable angina pectoris within the past 3 months
* Not pregnant or nursing and fertile patients must use barrier contraceptives

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2009-12-22 (Actual); Study Completion 2009-12-22 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) at each dose level | 22-28 days

SECONDARY OUTCOMES:
Safety measured by type, frequency and severity of adverse drug reactions | Every 4 weeks
  Safety measures by Common Terminology Criteria for Adverse Events (CTCAE)
Preliminary Efficacy od BGT226 | Every 8 weeks
  Measured by Response Evaluation criteria in Solid Tumors (RECIST)
Percent of patients in which an altered molecular status is detected for markers related to Pl3K signaling | Baseline, every 3 weeks
Biomarkers: Percentage of change, pre- versus post-treatment | Every month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kobe, Hyōgo